CLINICAL TRIAL: NCT05951075
Title: The Impact of Power Prenatal Supplements for Males on YO Score At-home Sperm Test Results Over a Three Month Course
Brief Title: Prospective Study on Power Prenatal Vitamins for Males on YO Score At-home Sperm Test Results
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Bird and Be Co Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BirdandBe
Record Dates: First submitted 2023-06-25; First posted 2023-07-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-08

CONDITIONS: Spermatogenesis and Semen Disorders; Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Count; Prenatal Care

STUDY DESIGN:
Intervention Model Description: Male patients that used the FDA approved YO Sperm at-home sperm analysis kit, and were identified with low YO Score results (20-40) will be recruited to take a 3 month course of supplements (Power Prenatal for Sperm), and a monthly YO Score at-home sperm test will be performed monthly for 3 consecutive months after starting the supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Power Prenatal for Sperm (Experimental): This is a single arm study. Participants will take supplements for 4 months. The supplements is Power Prenatal for Sperm (active ingredients - https://birdandbe.com/the-power-prenatal-for-sperm)
  Interventions: Dietary Supplement: Power Prenatal for Sperm

INTERVENTIONS:
Dietary Supplement: Power Prenatal for Sperm — A prenatal vitamin complex that includes numerous ingredients aim at improving sperm quality (ingredients: https://birdandbe.com/the-power-prenatal-for-sperm
  Other Names: Prenatal Vitamin

SUMMARY:
Male factor infertility is a leading cause of primary and secondary infertility. Poor sperm quality is defined as having an abnormal semen analysis.

There are now options to assess sperm quality with at-home sperm analysis kits, including an FDA approved Yo Sperm kit (https://yospermtest.com/) which analyzes the motile sperm concentration [concentration (millions / ml) x motility (Percentage motile)] and sperm quality (YO Score) which compares your results to laboratory standards and to other men who have fathered children.

The effects of supplements (vitamins, minerals, and anti-oxidants) on improving sperm quality are still debated. Taking additional supplements to improve sperm quality represent a modifiable risk-factor that would be an easy intervention for patients struggling with male factor infertility.

The life cycle of sperm production is estimated at 3 months, so any intervention would require a 3 month course to see its full effect.

The investigators hypothesize that a 90 day course of the "Power Prenatal for Sperm", a male fertility supplement by Bird&Be (https://birdandbe.com/the-power-prenatal-for-sperm) will improve sperm quality (YO Score) after taking the supplements.

DETAILED DESCRIPTION:
Male patients that used the FDA approved YO Sperm at-home sperm analysis kit, and were identified with a low YO Score result (20-40) will be potential candidates for this study.

An automated message about a potential research study for patients with a low YO Score results (20-40) will be sent to YO Sperm users. Interested participants will sign up to learn more about the research study. They will be prompted to complete further screening questions to ensure they're eligible study candidates (including inclusion and exclusion criteria, as well as primary residence country and province / state).

All study participants will be provided with IRB-approved study information materials and informed consent documents.

Once approved, and consented to participate, they will receive 3 months of The Power Prenatal for Males (https://birdandbe.com/collections/male-fertility/products/power-prenatal-vitamins-for-males) and re-evaluate the YO Score results monthly for 3 consecutive months after starting the supplements.

The monthly YO Scores will be compared between baseline, month 1, month 2 and month 3. YO Sperm's app will enable study participants to share results (YO Score) with the research team at each assessment. All data will be stored by the study sponsor in a secure and private manner compliant with HIPAA.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with at-home YO Sperm score between 20-40, corresponding to a MSC (motile sperm concentration) between 14-39 motile million / ml
* Ages 18-50
* Living in USA or Canada

Exclusion Criteria:

* Active smokers
* A known cause of male infertility (eg diagnosed varicocele, hormonal issue, history of testicular surgery, history of chemotherapy, etc)
* Not concurrently taking other forms of prenatal vitamins

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Focus on sperm quality
Enrollment: 174 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
YO Sperm Score | The YO Scores will be compared between baseline (prior to intervention) and after 3 months
  At-home YO Sperm score (10-90) YO Score is a ranking of a participants motile sperm concentration (MSC) compared to other men who have fathered children. The result is 10 to 90 in intervals of 10. A score of10 represents the lowest score (participant ranks above 10% of fathers), and 90 the highest score (participant ranks above 90% of fathers). The higher your YO Score, the more likely you are to achieve a pregnancy in a shorter amount of time. YO Score is a reliable tool for monitoring MSC changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nayot, BSc, MSc, MD, Principal Investigator — The Bird and Be Co Inc
Locations (1):
- Medical Electronic Systems, Encino, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salas-Huetos A, Rosique-Esteban N, Becerra-Tomas N, Vizmanos B, Bullo M, Salas-Salvado J. The Effect of Nutrients and Dietary Supplements on Sperm Quality Parameters: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Adv Nutr. 2018 Nov 1;9(6):833-848. doi: 10.1093/advances/nmy057. PMID 30462179
- See also: WHO laboratory manual for the examination and processing of human semen — https://www.who.int/publications/i/item/9789240030787